CLINICAL TRIAL: NCT06605885
Title: An Observational, Prospective, Multicenter Study to Evaluate the Biologic Use and Outcomes in Chinese Asthma Patients
Acronym: PRESENTII
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00039
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter, observational, prospective study to evaluate the asthma biologic use features and clinical outcomes in China. Patients will undergo clinical assessments and receive standard medical care as determined by the treating physician.

DETAILED DESCRIPTION:
This study is a multicenter, observational, prospective study to evaluate the asthma biologic use features and clinical outcomes in China. Patients will undergo clinical assessments and receive standard medical care as determined by the treating physician.

Approximately 200 patients with a physician diagnosis of asthma and prescribed with asthma biologics at visit 1 will be enrolled in this study, distributed among 50 sites across different regions in China.

During the study period, patients will be identified consecutively and, if they meet eligibility criteria and provide informed consent will be entered into this observational study. Patients should have an asthma diagnosis and be prescribed at least once with biologics for asthma treatment at enrollment (Visit 1, Week 0).

After the enrollment, subjects will be followed up at Visit 2(Week 24) and Visit 3 (Week 52). V1, V2 and V3 will be followed up by on-site visit. At Visit 1, data within last 12 months will be retrospectively collected as baseline. Patients existing medical record (MR) data will be collected in week 24 and week 52. PROs (Asthma control test [ACT], Asthma Quality of Life Questionnaire (+12) [AQLQ(S)+12]) should be performed at Visit 1, Visit 2 and Visit 3.

No additional mandated interventions on top of routinely performed physician visits, examinations or treatments will be required. Patients will not receive any experimental disease management intervention or experimental treatment as a result of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese, Female or Male
2. Age: no limitation
3. Physician-confirmed asthma diagnosis with documented evidence of diagnosis or evidence of variable expiratory airflow limitation (e.g., from bronchodilator reversibility testing or other tests).
4. Participants or their legal guardians must be able to provide informed consent.
5. Prescription of asthma biologics at enrolment.

   Exclusion Criteria:
6. Participation in an interventional study within the last 3 months.
7. Any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study with the usage of biologics, or may influence the results of the study, or the patient's ability to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 200 asthma patients will be enrolled in this study distributed among 50 sites in China.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of days covered (PDC) with asthma biologics during 52 weeks | week52
  to describe the persistence to asthma biologics using proportion of days covered (PDC) with asthma biologics during 52 weeks.

SECONDARY OUTCOMES:
Time from asthma onset to first biologic initiation(month) | week0
  To describe asthma biologics treatment features
Duration (days) of treatment with different type of biologics. | week 52
  To describe asthma biologics treatment features
Proportion of patients discontinued biologics in week 24 and week 52. | week24,week52
  To describe asthma biologics treatment features
Proportion of participants switching to other biologics for asthma in week 24 and week 52. | week24,week52
  To describe asthma biologics treatment features
Proportion of participants with concurrent used of multiple biologics in week 24 and week 52. | week24,week52
  To describe asthma biologics treatment features
Proportion of different categories including anti-IL5, anti-IL5R, anti-IL4R, anti-IgE and anti-TSLP of biologics during 52 weeks | week 52
  To describe asthma biologics treatment features
Proportion of patients experiencing asthma related hospitalizations during 52 weeks | week 52
  To describe effect of biologics on healthcare care resource utilization (HCRU)
Cost of asthma related hospitalization during 52 weeks | week 52
  To describe effect of biologics on healthcare care resource utilization (HCRU)
Days on asthma related sick leaves during 52 weeks | week 52
  To describe effect of biologics on healthcare care resource utilization (HCRU)
Number of emergency visit during 52 weeks | week 52
  To describe effect of biologics on healthcare care resource utilization (HCRU)
Annualized exacerbation rates over 52 weeks | week 52
  To describe clinical outcomes of biologics including lung function, exacerbation, symptom control and quality of life in two subgroups
Change from baseline of FEV1 at week 24, 52 | week0,week 24, week 52
  To describe clinical outcomes of biologics including lung function, exacerbation, symptom control and quality of life in two subgroups
Change from baseline of ACT score at week 24, 52 | week0,week 24,week52
  To describe clinical outcomes of biologics including lung function, exacerbation, symptom control and quality of life in two subgroups
Change from baseline of AQLQ(S)+12 score at week 24, 52 | week0,week24,week52
  To describe clinical outcomes of biologics including lung function, exacerbation, symptom control and quality of life in two subgroups
Change of proportion of patients with high-dosage ICS from baseline to week 24,52 | week0,week24,week52
  To describe maintenance treatment change after biologic initiation in two subgroups
Change of proportion of patients with maintenance OCS from baseline to week 24,52 | week0,week 24,Week 52
  To describe maintenance treatment change after biologic initiation in two subgroups
Proportion of days covered (PDC) with maintenance medication at baseline (in last 3 months) | week0
  To describe the characteristics including background therapy, biomarkers, asthma triggers and comorbidities of biologics treated asthma patients in two subgroups
Levels of bEOS at baseline | week0
  To describe the characteristics including background therapy, biomarkers, asthma triggers and comorbidities of biologics treated asthma patients in two subgroups
Levels of FeNO at baseline | week0
  To describe the characteristics including background therapy, biomarkers, asthma triggers and comorbidities of biologics treated asthma patients in two subgroups
Levels of IgE at baseline | week0
  To describe the characteristics including background therapy, biomarkers, asthma triggers and comorbidities of biologics treated asthma patients in two subgroups

OTHER OUTCOMES:
Proportion of different reasons for biologics discontinuation | week52
  To describe reasons for biologic discontinuation and switching, including asthma control, adverse event, cost or other more reasons.
Proportion of different reasons for biologics switching | week52
  To describe reasons for biologic discontinuation and switching, including asthma control, adverse event, cost or other more reasons.
Incidence of all AEs and SAEs | week52
  To describe reasons for biologic discontinuation and switching, including asthma control, adverse event, cost or other more reasons.

CONTACTS AND LOCATIONS:
Overall Officials: YuBiao Guo, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University
Locations (30):
- China (30):
  - Research Site, Hohhot, China
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Quanzhou
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. 'Yes' , indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/